CLINICAL TRIAL: NCT05556291
Title: Efficacy, Safety & Tolerability of Combination of Ertugliflozin and Sitagliptin in Patients With Type II Diabetes Mellitus
Brief Title: Combination of Ertugliflozin And Sitagliptin Efficacy, Safety & Tolerability (CEASE Diabetes) Study
Acronym: CEASE
Status: Completed | Type: Observational
Sponsor: Getz Pharma (Industry)
Collaborators: Primary Care Diabetes Association, Pakistan (Other)
Responsible Party: Sponsor
Other Study IDs: GTZ-DM-006-22
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Efficacy; Safety; Tolerability
Keywords: Efficacy, Safety, Tolerability, Ertugliflozin, Sitgliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Combinations of Oral Blood Glucose Lowering Drugs — Combination of Ertugliflozin and Sitagliptin

SUMMARY:
Open-label, prospective, observational, single arm, multi-center, post-marketing surveillance study to evaluate the efficacy, safety and tolerability of Ertugliflozin and Sitagliptin Con-initiation in patients with Type II Diabetes Mellitus in the Pakistani population. The study duration will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic males & females between 18-65 years.
* HbA1c: 7.0% - 10.0%
* Patient uncontrolled on oral anti-diabetics and lifestyle modifications for at least 3 months.
* eGFR >60 mL/min/1.73m2.
* Patient who will give informed consent
* Patient who are SGLT2i naïve

Exclusion Criteria:

* History of severe hypoglycemia for the last three months (<70mg/dL)
* Pregnant or lactating females
* History of renal and/or hepatic dysfunctions, where RFT and Urine R/E is abnormal
* History of recurrent urinary tract infection (UTI) and/or past 3 months' history of UTI and its treatment
* Patients who have been admitted to the hospital in the past 3 months for diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic state.
* History of acute coronary syndrome or myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack.
* History of active liver disease, including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Patient with diabetic foot ulcers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic uncontrolled on lifestyle modification and OADs
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c% to the last-observation. | up to 24 weeks
  Efficacy
Change from baseline in fasting plasma glucose to the last- observation on treatment | 24 weeks
  Efficacy
Change from baseline in bodyweight & BMI | till 24 weeks
  Efficacy

SECONDARY OUTCOMES:
Frequency of adverse events during the course of study follow-up | 24 weeks
  Safety
Frequency of serious adverse events | up to 24 weeks
  Safety
Percentage of patients who discontinued investigational drug due to adverse events | up to 24 weeks
  Tolerability

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Doctor's Plaza, Karachi, Sindh
  - Khan's Clinic, Karachi, Sindh
  - PECHS, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Diabetes Federation. IDF Diabetes Atlas, 10th edn.: International Diabetes Federation, 2021. http://www.diabetesatlas.org
- [Background] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Background] Aamir AH, Ul-Haq Z, Mahar SA, Qureshi FM, Ahmad I, Jawa A, Sheikh A, Raza A, Fazid S, Jadoon Z, Ishtiaq O, Safdar N, Afridi H, Heald AH. Diabetes Prevalence Survey of Pakistan (DPS-PAK): prevalence of type 2 diabetes mellitus and prediabetes using HbA1c: a population-based survey from Pakistan. BMJ Open. 2019 Feb 21;9(2):e025300. doi: 10.1136/bmjopen-2018-025300. PMID 30796126
- [Background] Lin X, Xu Y, Pan X, Xu J, Ding Y, Sun X, Song X, Ren Y, Shan PF. Global, regional, and national burden and trend of diabetes in 195 countries and territories: an analysis from 1990 to 2025. Sci Rep. 2020 Sep 8;10(1):14790. doi: 10.1038/s41598-020-71908-9. PMID 32901098
- [Background] van Baar MJB, van Ruiten CC, Muskiet MHA, van Bloemendaal L, IJzerman RG, van Raalte DH. SGLT2 Inhibitors in Combination Therapy: From Mechanisms to Clinical Considerations in Type 2 Diabetes Management. Diabetes Care. 2018 Aug;41(8):1543-1556. doi: 10.2337/dc18-0588. PMID 30030256
- [Background] Verbrugge FH. Role of SGLT2 Inhibitors in Patients with Diabetes Mellitus and Heart Failure. Curr Heart Fail Rep. 2017 Aug;14(4):275-283. doi: 10.1007/s11897-017-0340-1. PMID 28647919
- [Background] Mazidi M, Rezaie P, Gao HK, Kengne AP. Effect of Sodium-Glucose Cotransport-2 Inhibitors on Blood Pressure in People With Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis of 43 Randomized Control Trials With 22 528 Patients. J Am Heart Assoc. 2017 May 25;6(6):e004007. doi: 10.1161/JAHA.116.004007. PMID 28546454
- [Background] Scott R, Loeys T, Davies MJ, Engel SS; Sitagliptin Study 801 Group. Efficacy and safety of sitagliptin when added to ongoing metformin therapy in patients with type 2 diabetes. Diabetes Obes Metab. 2008 Sep;10(10):959-69. doi: 10.1111/j.1463-1326.2007.00839.x. Epub 2008 Jan 14. PMID 18201203
- [Background] Chung WK, Erion K, Florez JC, Hattersley AT, Hivert MF, Lee CG, McCarthy MI, Nolan JJ, Norris JM, Pearson ER, Philipson L, McElvaine AT, Cefalu WT, Rich SS, Franks PW. Precision Medicine in Diabetes: A Consensus Report From the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2020 Jul;43(7):1617-1635. doi: 10.2337/dci20-0022. PMID 32561617
- [Background] McNeill AM, Davies G, Kruger E, Kowal S, Reason T, Ejzykowicz F, Hannachi H, Cater N, McLeod E. Ertugliflozin Compared to Other Anti-hyperglycemic Agents as Monotherapy and Add-on Therapy in Type 2 Diabetes: A Systematic Literature Review and Network Meta-Analysis. Diabetes Ther. 2019 Apr;10(2):473-491. doi: 10.1007/s13300-019-0566-x. Epub 2019 Jan 28. PMID 30689140
- [Background] Shankar RR, Zeitler P, Deeb A, Jalaludin MY, Garcia R, Newfield RS, Samoilova Y, Rosario CA, Shehadeh N, Saha CK, Zhang Y, Zilli M, Scherer LW, Lam RLH, Golm GT, Engel SS, Kaufman KD. A randomized clinical trial of the efficacy and safety of sitagliptin as initial oral therapy in youth with type 2 diabetes. Pediatr Diabetes. 2022 Mar;23(2):173-182. doi: 10.1111/pedi.13279. Epub 2021 Dec 22. PMID 34779087
- [Background] Miller S, Krumins T, Zhou H, Huyck S, Johnson J, Golm G, Terra SG, Mancuso JP, Engel SS, Lauring B. Ertugliflozin and Sitagliptin Co-initiation in Patients with Type 2 Diabetes: The VERTIS SITA Randomized Study. Diabetes Ther. 2018 Feb;9(1):253-268. doi: 10.1007/s13300-017-0358-0. Epub 2018 Jan 8. PMID 29313282
- [Background] Pratley RE, Eldor R, Raji A, Golm G, Huyck SB, Qiu Y, Sunga S, Johnson J, Terra SG, Mancuso JP, Engel SS, Lauring B. Ertugliflozin plus sitagliptin versus either individual agent over 52 weeks in patients with type 2 diabetes mellitus inadequately controlled with metformin: The VERTIS FACTORIAL randomized trial. Diabetes Obes Metab. 2018 May;20(5):1111-1120. doi: 10.1111/dom.13194. Epub 2018 Jan 25. PMID 29266675
- See also: International Diabetes Federation. IDF Diabetes Atlas, 10th edn.: International Diabetes Federation, 2021. — http://www.diabetesatlas.org